CLINICAL TRIAL: NCT06827483
Title: Identifying Asymmetries in Reaction Time and Reach Distance by Adding a Neurocognitive Component to the Y-Balance Test of the Lower Quarter
Brief Title: Adding Neurocognitive Component to Balance Test
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00117009
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; Y-Balance Test; Reaction Time; Return to Sport
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals: Healthy individuals without a history of ACL injury or reconstruction
  Interventions: Other: Neurocognitive Component
- ACL (anterior cruciate ligament) reconstruction patients: Patients who have undergone ACL reconstruction and present for performance testing to measure readiness for sport participation
  Interventions: Other: Neurocognitive Component

INTERVENTIONS:
Other: Neurocognitive Component — A neurocognitive component will be added to the Y Balance Test

SUMMARY:
By introducing BlazePods as a neurocognitive addition to the YBT, this study aims to determine whether this addition impacts balance performance and/or reach distances between the operative and non-operative limbs of patients recovering from ACL reconstruction. Findings will contribute to optimizing return-to-sport protocols and enhancing late-stage rehabilitation program designs.

DETAILED DESCRIPTION:
The study team will measure performance under two conditions: the standard Y-Balance Test (YBT) and the YBT with an added neurocognitive component (YBT+NC). For the YBT+NC, the study team will attach Blaze Pods to the target area of the three reach indictors: anterior (A), posteromedial (PM), and posterolateral (PL). The Blaze Pods will light up in random sequences, requiring participants to slide the illuminated reach indicator as far as possible while maintaining balance on the stationary stance limb. Reaction time, individual reach distances (PM,PL,A), YBT composite score, and number of errors will be recorded and compared bilaterally.

To first establish feasibility and clinical utility, a pilot group of healthy participants will perform both the YBT and the YBT+NC with two simultaneous testers on two separate occasions separated by at least one day but no more than 28 days. The differences in reach distances, composite scores, and reaction times between the two test conditions will be compared. The study team will also determine intra- and inter-rater reliability as well as any learning effects.

For the patient cohort, the study team will employ a cross-sectional design to measure patients presenting for physical performance testing battery between 5-8 months post-anterior cruciate ligament reconstruction/repair (ACLR). This visit is standard of care for this population. If the patient is able to pass the initial screening test (maintain pain-free single leg balance for 10 seconds) a physical therapist will have the patient perform both the YBT and the YBT+NC as described above. The study team will compare the side-to-side differences between reaction time, reach distance, and number of errors (loss of balance) made.

ELIGIBILITY:
Inclusion Criteria:

* All participants: 18-25 years old
* All participants: MARX activity questionnaire of greater than 10
* All participants: able to follow verbal instructions
* For patient participants: ACL Repair or Reconstruction within past 5-7 months

Exclusion Criteria:

* Healthy participants: Chronic Ankle Instability
* Healthy participants: Prior lower extremity surgery
* Healthy participants: LE injury <6 months ago
* Healthy participants: current LE pain
* Healthy participants: visual deficits
* Healthy participants: vestibular or neurological deficits affecting balance
* Healthy participants: unable to maintain single leg stance for 10 seconds
* Healthy participants: unable to read or speak English
* For patient participants: Chronic Ankle Instability
* For patient participants: current LE pain
* For patient participants: multi-ligament procedure
* For patient participants: prior surgery on uninvolved limb
* For patient participants: visual deficits
* For patient participants: vestibular or neurological deficits affecting balance
* For patient participants: unable to read or speak English
* For patient participants: unable to maintain single leg stance for 10 seconds

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants will be recruited from the community. Patient participants will be recruited from the study center's population of patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Y-Balance Test - reach distance with and without neurocognitive component | Day 1
  Reach Distances and Composite Score compared between left and right sides.
Y-Balance Test - composite score with and without neurocognitive component | Day 1
  Composite Score compared between left and right sides.
Reaction Time Asymmetry between limbs | Day 1
  Difference in reaction time between limbs

SECONDARY OUTCOMES:
Reliability of Y-Balance Test - Inter-rater | Day 8
  Reliability of Y-Balance Test - Inter-rater
Reliability of Y-Balance Test - Intra-rater | Day 8
  Reliability of Y-Balance Test - Intra-rater
Reliability of Reaction Time Measurements - Inter-rater | Day 8
  Reliability of Reaction Time Measurements - Inter-rater
Reliability of Reaction Time Measurements - Intra-rater | Day 8
  Reliability of Reaction Time Measurements - Intra-rater

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tisherman, MD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No